CLINICAL TRIAL: NCT04945603
Title: Poor Grade Aneurysmal Subarachnoid Hemorrhage Multicentric Study Group
Brief Title: Poor Grade Aneurysmal Subarachnoid Hemorrhage Study Group
Acronym: POGASH
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); A.O. Ospedale Papa Giovanni XXIII (Other); ASL Taranto (Other); Ospedale V. Fazzi (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Pietro Panni, Principal Investigator, IRCCS San Raffaele
Other Study IDs: POGASH
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Poor Grade Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Poor Grade Subarachnoid Hemorrhage: All patients (prospective and retrospective) included will have to present a subarachnoid hemorrhage defined poor grade according to the WFNS scale due to the rupture of an intracranial aneurysm.
  The patients are managed according to both most recent international guidelines on the specific disease (Stroke, May 2012) and according to national and institutional guidelines/protocols.
  Interventions: Other: Standard management according to international/national guidelines

INTERVENTIONS:
Other: Standard management according to international/national guidelines — Standard management according to international/national guidelines. Observational study

SUMMARY:
Multicentric registry study in order to define outcome, predictors, treatment effects and their modifiers in poor grade aneurysmal subarachnoid haemorrhage patients.

The search for outcome predictors is going to be subdivided into three main research areas:

1. outcome predictors in the emergency department (so called "early brain injury phase").
2. outcome predictors in the neurocritical care unit (so called "delayed brain injury phase").
3. Treatment strategies. Two other areas of research are identified: delayed cerebral ischemia (incidence, treatment, predictors, impact on outcome) and long term follow-up (recent evidences suggest that there may be a non-negligible proportion of poor grade subarachnoid hemorrhage patients who may benefit from substantial improvement at long-term (after 6-12 months of follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department because of aneurysmal subarachnoid hemorrhage of poor grade (IV-V) according to the WFNS classification.

Exclusion Criteria:

* Patients younger than 18 years old.
* Pregnant or breast-feeding patients.
* Aneurysmal subarachnoid hemorrhage due to trauma or vascular malformations other than cerebral aneurysms.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to the emergency department because of aneurysmal subarachnoid hemorrhage of poor grade (IV-V) according to the WFNS classification
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome | 6 months.
  modified Rankin Scale
Clinical Outcome | 12 months
  modified Rankin Scale (mRS). Scale ranging from 0 (no symptoms) to 6 (dead) with higher scores indicating increasing neurological disability.

SECONDARY OUTCOMES:
Long-Term clinical outcome | 12-60 months
  modified Rankin Scale (mRS). Scale ranging from 0 (no symptoms) to 6 (dead)
Delayed Cerebral Ischemia | onset-30 days
  Delayed Cerebral Ischemia
Rebleeding | onset-48hours
  Rebleeding
Treatment Complications | onset-1 week
  Treatment Complications
Decompressive Craniotomy | onset-3 weeks
  Incidence, strategy (primary or secondary), predictors and clinical impact
Ventriculo-peritoneal shunt | onset-4 weeks
  Incidence, strategy (primary or secondary), predictors and clinical impact
CSF drainage | onset-3 weeks
  Use of external ventricular drainage or lumbar drainage according to institutional protocol. Clinical impact.
Volumetric analysis of intracranial bleeding | onset-24hours
  Volumetric analysis and distribution assessment of intracranial bleeding. Clinical impact
Volumetric analysis of delayed cerebral ischemia | onset-3 weeks
  Volumetric analysis and location assessment of delayed cerebral ischemia. Clinical impact

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Panni, P.I., M.D., Principal Investigator — Department of Neuroradiology, Department of Neurosurgery
Locations (10):
- Italy (10):
  - ASST Ospedale Papa Giovanni XXIII, Bergamo
  - IRCCS Bellaria, Bologna
  - Azienda Ospedaliera Spedali Civili, Brescia
  - Ospedale Vito Fazzi, Lecce
  - IRCCS San Raffaele, Milan
  - Ospedale Maggiore della Città di Novara, Novara
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Santissima Annunziata, Taranto
  - Azienda Ospedaliera Universitaria Integrata, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panni P, Ambrosi A; POGASH (Poor Grade Aneurysmal Subarachnoid Hemorrhage) Investigators. In Reply: Clinical Impact and Predictors of Aneurysmal Rebleeding in Poor-Grade Subarachnoid Hemorrhage: Results From the National POGASH Registry. Neurosurgery. 2023 Dec 1;93(6):e174-e176. doi: 10.1227/neu.0000000000002691. Epub 2023 Sep 21. No abstract available. PMID 37732736
- [Result] Panni P, Riccio L, Cao R, Pedicelli A, Marchese E, Caricato A, Feletti A, Testa M, Zanatta P, Gitti N, Piva S, Mardighian D, Semeraro V, Nardin G, Lozupone E, Paiano G, Picetti E, Montanaro V, Petranca M, Bortolotti C, Scibilia A, Cirillo L, Lanterna AL, Ambrosi A, Mortini P, Beretta L, Falini A. Clinical Impact and Predictors of Aneurysmal Rebleeding in Poor-Grade Subarachnoid Hemorrhage: Results From the National POGASH Registry. Neurosurgery. 2023 Sep 1;93(3):636-645. doi: 10.1227/neu.0000000000002467. Epub 2023 Apr 3. PMID 37010298